CLINICAL TRIAL: NCT04831086
Title: To Optimize Antenatal Management of Women Admitted With Pre Term Labor and Intact Membranes Using Multivariable Prediction Models: Multicenter Randomised Control Trial (OPTIM-PTL)
Brief Title: To Optimize Antenatal Management of Women With Pre Term Labor Using Amniocentesis
Acronym: OPTIM-PTL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Hospital Vall d'Hebron (Other); Hospital Universitario La Fe (Other); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other); Consorci Sanitari de Terrassa (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Universitario Puerta del Mar (Other); Hospital Sant Joan de Deu (Other); Germans Trias i Pujol Hospital (Other); University Hospital Virgen de las Nieves (Other); Hospital Clínico Universitario Lozano Blesa (Other); Parc Taulí Hospital Universitari (Other); Complexo Hospitalario Universitario de A Coruña (Other); Hospital Son Llatzer (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital Universitario de Torrejón (Unknown)
Responsible Party: Principal Investigator, Teresa Cobo Cobo, Senior Specialist, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIM-PTL
Record Dates: First submitted 2021-03-24; First posted 2021-04-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Preterm Birth; Preterm Labor; Intra-amniotic Infection; Amniocentesis Affecting Fetus or Newborn
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Tocolytic Agents

STUDY DESIGN:
Intervention Model Description: Pregnant women with singleton pregnancies admitted with a diagnosis of preterm labor and intact membranes between 23.0 and 34.6 weeks, not in labor at randomization and who do not meet exclusion criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): In the intervention arm, the management will be optimized according to the risk of the predictive model. The predictive model of intra-amniotic infection includes maternal C-reactive protein (CRP) (in mg/L) and amniotic fluid glucose (in mg/dL), and the predictive model of spontaneous preterm delivery within 7 days includes gestational age (in weeks), cervical length (in mm), amniotic fluid glucose (in mg/dL) and Interleukin (IL)-6 (in a log10 scale). High risk will be defined when the risk is > 10% in the predictive model of spontaneous delivery in 7 days and > 20% in the predictive model of intra-amniotic infection:
  1. If low-risk: we will optimize the standard management reducing the dose of steroids (e.g not administering second doses), tocolysis duration and facilitating discharge home.
  2. If high-risk: we will follow the standard management of each center and we will treat with antibiotics
  Interventions: Drug: Steroid Drug; Drug: Tocolytic Agents
- Control (No Intervention): In the control arm the standard management of each center will be followed regarding doses of steroids, duration of tocolysis or maternal stay length duration.

INTERVENTIONS:
Drug: Steroid Drug — Steroids doses will be optimized in the intervention group according the risk based on predictive models
  Arms: Intervention
Drug: Tocolytic Agents — Tocolysis duration will be optimized in the intervention group according the risk based on predictive models
  Arms: Intervention

SUMMARY:
Implementation of prediction models of risk of spontaneous delivery within 7 days or of intra-amniotic infection in women with preterm labor and intact membranes

DETAILED DESCRIPTION:
To evaluate whether the implementation of prediction models of risk of spontaneous delivery within 7 days or of intra-amniotic infection:

1. Optimises antenatal management (regarding steroids, tocolysis, antibiotics, maternal length stay duration) without worsening perinatal outcomes.
2. It is a cost-effective strategy.
3. It improves neonatal outcome (in premature newborns <30 weeks), and reduces infectious maternal morbility.
4. It improves neurodevelopmental outcome at 1.2 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton pregnancies admitted with a diagnosis of preterm labor between 23.0 and 34.6 weeks, not in labor at randomization and who do not meet exclusion criteria.

Exclusion Criteria:

* Women who do no accept to be part of the study
* Maternal age < 18 years
* Multiple gestations
* Clinical chorioamnionitis at randomization (defined by the presence of fever above 38 celsius degrees (ºC), fetal tachycardia (>160 heart beat per minute >10 minutes), maternal White blood cells > 15000/mm3 (not justified by the administration of antenatal steroids).
* Cervical dilatation > 3 cm
* Major structural malformations of fetal complications that are related to neurodevelopmental impairment.
* Technical problems to perform an amniocentesis (prediction models include information from amniotic fluid: glucose and IL-6 concentration).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Antenatal steroid doses | through study completion, an average of 1 year
  Number of antenatal steroid doses administered

SECONDARY OUTCOMES:
maternal stay length | through study completion, an average of 1 year
  Maternal length of hospital stay (in days).
Clinical chorioamnionitis | through study completion, an average of 1 year
  Clinical chorioamnionitis occurrence defined by the presence of maternal fever >=38ºC, fetal tachycardia > 160 bpm, leukocytes > 14000/m2 without steroids effect and cervical purulent fluid

OTHER OUTCOMES:
Tocolysis duration | through study completion, an average of 1 year
  Tocolysis duration (in days)
Gestational age at delivery | through study completion, an average of 1 year
  Gestational age at delivery
Spontaneous delivery within 7 days after admission | through study completion, an average of 1 year
  Spontaneous delivery within 7 days after admission (yes/no),
Microbial invasion of amniotic cavity | through study completion, an average of 1 year
  Microbial invasion of amniotic cavity (yes/no) defined by the presence of a positive amniotic fluid culture, detection of 16S rRNA gene or visualization of microorganisms at the Gram stain
Cost analyses | through study completion, an average of 1 year
  Cost analyses: The following resource items will be collected: maternal and neonatal admissions, method of delivery, type of induction, outpatient visits, emergency visits, medication, surgical procedures, maternal stay length.
Maternal morbidity | through study completion, an average of 1 year
  Maternal morbidity (yes/no) including intrapartum fever, endometritis, infection of surgical wound, sepsis, curettage, admission to ICU, hysterectomy, need for transfusion, maternal death.
Neonatal length of hospital stay | through study completion, an average of 1 year
  Neonatal length of hospital stay (days)
Neonatal birthweight (in grams) | through study completion, an average of 1 year
  Neonatal anthropometric measurements
height (in centimeters) | through study completion, an average of 1 year
  Neonatal anthropometric measurements
cephalic, thoracic and abdominal perimeters (in millimeters) | through study completion, an average of 1 year
  Neonatal anthropometric measurements
arm circumference (in centimeters) | through study completion, an average of 1 year
  Neonatal anthropometric measurements
Adverse neonatal outcome | through study completion, an average of 1 year
  A composite adverse neonatal outcome (yes/no) defined as the presence or one or more of the following outcomes: fetal or neonatal death, early onset sepsis, moderate/severe bronchopulmonary dysplasia, severe intraventricular haemorrhage, periventricular leukomalacia, surgical necrotizing enterocolitis, retinopathy requiring laser treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Cobo, MD, PhD, Principal Investigator — Fundació Recerca Biomèdica Clínica
Locations (1):
- Fundació Recerca Biomèdica Clínica, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after the end of the study
Access Criteria: https://apps.sjdhospitalbarcelona.org/redcap/

REFERENCES:
- [Result] Cobo T, Aldecoa V, Figueras F, Herranz A, Ferrero S, Izquierdo M, Murillo C, Amoedo R, Rueda C, Bosch J, Martinez-Portilla RJ, Gratacos E, Palacio M. Development and validation of a multivariable prediction model of spontaneous preterm delivery and microbial invasion of the amniotic cavity in women with preterm labor. Am J Obstet Gynecol. 2020 Sep;223(3):421.e1-421.e14. doi: 10.1016/j.ajog.2020.02.049. Epub 2020 Mar 5. PMID 32147290
- [Derived] Cobo T, Aldecoa V, Bartha JL, Bugatto F, Paz Carrillo-Badillo M, Comas C, Diago-Almeda V, Ferrero S, Goya M, Herraiz I, Marti-Malgosa L, Olivella A, Paules C, Vives A, Figueras F, Palacio M, Gratacos E; OPTIM-PTL group. Assessment of an intervention to optimise antenatal management of women admitted with preterm labour and intact membranes using amniocentesis-based predictive risk models: study protocol for a randomised controlled trial (OPTIM-PTL Study). BMJ Open. 2021 Sep 28;11(9):e054711. doi: 10.1136/bmjopen-2021-054711. PMID 34588268
- See also: Predictive models of spontaneous delivery within 7 days and of intra-amniotic infections description — https://doi.org/10.1016/j.ajog.2020.02.049

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT04831086/Prot_SAP_000.pdf